CLINICAL TRIAL: NCT01025466
Title: A Multicenter, Randomized, Open-label Study to Compare the Tolerability Between Rivastigmine Patch Monotherapy and Combination Therapy With Memantine in Patients With Alzheimer's Disease
Brief Title: Exelon Patch and Combination With Memantine Comparative Trial
Acronym: EXPECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Seong Hye Choi, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXPECT
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rivastigmine patch monotherapy (Active Comparator)
  Interventions: Drug: Rivastigmine transdermal patch
- Combination therapy with memantine (Active Comparator)
  Interventions: Drug: Rivastigmine transdermal patch (Exelon patch), memantine

INTERVENTIONS:
Drug: Rivastigmine transdermal patch (Exelon patch), memantine — All patients start on a 5-cm2 rivastigmine patch and their dose is increased to a 10-cm2 patch after 4 weeks. Patients will be randomly allocated to 1 of 2 treatment groups of rivastigmine patch monotherapy and combination therapy with memantine at the baseline visit (week 9)and treated with the drugs for 16 weeks.
  Other Names: exelon patch, ebixa
  Arms: Combination therapy with memantine
Drug: Rivastigmine transdermal patch — All patients start on a 5-cm2 rivastigmine patch and their dose is increased to a 10-cm2 patch after 4 weeks. Patients will be randomly allocated to 1 of 2 treatment groups of rivastigmine patch monotherapy and combination therapy with memantine at the baseline visit (week 9)and treated with the drugs for 16 weeks.
  Other Names: exelon patch
  Arms: rivastigmine patch monotherapy

SUMMARY:
The primary objective is to compare the tolerability between rivastigmine patch monotherapy and combination therapy with memantine in patients with Alzheimer's disease (AD). The secondary objective is to compare the efficacy and safety between rivastigmine patch monotherapy and combination therapy with memantine in patients with AD. The study hypothesis is that the tolerability of the combination therapy with memantine is not inferior to that of rivastigmine patch monotherapy in AD patients.

DETAILED DESCRIPTION:
Recently, the rivastigmine patch demonstrated efficacy comparable to the highest doses of rivastigmine capsules, with markedly improved tolerability profile. We hypothesized that combination of memantine and rivastigmine patch will be safe and well tolerated and result in more clinical benefit in patients with AD in comparison with rivastigmine patch monotherapy, for the mechanisms of the drugs are different.

ELIGIBILITY:
Inclusion Criteria:

* Dementia by DSM-IV and probable AD by NINCDS-ADRDA
* Age of 50 to 90 years
* Mini-Mental State Examination (MMSE) score of 10 to 20
* Brain MRI or CT scan consistent with a diagnosis of probable AD
* The caregiver must meet the patient at least once a week and be sufficiently familiar with the patient to provide accurate data.
* Ambulatory or ambulatory-aided (is, walker or cane) ability
* Written informed consent will be obtained from the patient (if possible) and from the patient's legally acceptable representative. Even if unable to provide written informed consent, the patient must assent verbally to participating in the study.

Exclusion Criteria:

* Patients with evidence of severe or unstable physical illness, i.e., acute and severe asthmatic conditions, severe or unstable cardiovascular disease, active peptic ulcer disease, severe hepatic or renal disease, or any medical condition which would prohibit them from completing the study
* Any psychiatric or primary neurodegenerative disorder other than AD
* Any patients with hearing or visual problem that can disturb the efficient evaluation of the patients.
* Any patients with a history of drug addiction or alcohol addiction for the past 10 years
* Patients with bradycardia (bpm less than 50) or sick sinus syndrome or conduction defects (sino-atrial block, second ot third degree A-V blocks
* Clinically significant laboratory abnormalities to affect cognitive function (i.e.abnormal thyroid function test, abnormal low level of vitamin B12 or folate, or syphilis, etc)
* History of allergy to topical products containing any of the constitution of the patches
* Current diagnosis of an active skin lesion
* Involved in other clinical trials or treated by experimental drug within 4 weeks
* Patients with hypersensitivity to cholinesterase inhibitors

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Retention rate at week 16 after randomization | End point (16 weeks after randomization)

SECONDARY OUTCOMES:
Change from baseline at week 16 in Alzheimer's Disease Assessment Scale-Cognitive subscale | 16 weeks after randomization
Change from baseline at week 16 in Mini-Mental State Examination | 16 weeks after randomization
Change from baseline at week 16 in Frontal Assessment Battery | 16 weeks after randomization
Change from baseline at week 16 in Alzheimer's Disease Cooperative Study - Activities of Daily Living | 16 weeks after randomization
Change from baseline at week 16 in Caregiver-Administered Neuropsychiatric Inventory | 16 weeks after randomization
Change from baseline at week 16 in Cohen Mansfield Agitation Inventory | 16 weeks after randomization
Change from baseline at week 16 in Clinical Dementia Rating Scale-Sum of Boxes | 16 weeks after randomization
Safety | from baseline to end-point

CONTACTS AND LOCATIONS:
Overall Officials: Seong Choi, MD, Principal Investigator — Department of Neurology, Inha University Hospital
Locations (26):
- South Korea (26):
  - Soonchunhyang University Hospital, Bucheon-si
  - The Catholic University of Korea Hospital, Bucheon-si
  - Donga University Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Keimyung University Dongsan Medical Center, Daegu
  - Daejun Eulji University Hopistal, Daejun
  - Dongguk University Medical Center, Goyang
  - Myongji Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Inha Univeristy Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Pusan National University Hospital, Pusan
  - Maryknoll Hospital, Pusan
  - Bobath Memorial Hospital, Seongnam
  - Kyughee University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Sungkyunkwan University, Samsung Seoul Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Hallym University Hospital, Seoul
  - Ewha Womans University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul Eulji Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Choi SH, Park KW, Na DL, Han HJ, Kim EJ, Shim YS, Lee JH; Expect Study Group. Tolerability and efficacy of memantine add-on therapy to rivastigmine transdermal patches in mild to moderate Alzheimer's disease: a multicenter, randomized, open-label, parallel-group study. Curr Med Res Opin. 2011 Jul;27(7):1375-83. doi: 10.1185/03007995.2011.582484. Epub 2011 May 12. PMID 21561398